CLINICAL TRIAL: NCT05025189
Title: Effect of Grape Consumption on the Microbiome in Healthy Subjects: A Pilot Study
Brief Title: The Effect of Grape Consumption on Increasing the Good Bacteria in the Human Intestine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The California Table grape Commission (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Chief, Division of Clinical Nutrition, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-001635
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This will be a two phase intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Table Grape (Active Comparator): Subjects will consume 4 weeks of (two servings) of standardized Freeze-Dried Whole Table Grape Powder
  Interventions: Other: Table Grape Powder
- Beige Diet (Placebo Comparator): Subjects will consume 4 weeks of a beige diet (low in fiber and low in polyphenols)
  Interventions: Other: Beige Diet

INTERVENTIONS:
Other: Table Grape Powder — Freeze Dried Whole Table Grape Powder
  Arms: Table Grape
Other: Beige Diet — Low Fiber, low polyphenol Diet
  Arms: Beige Diet

SUMMARY:
This pilot study will assess the ability of daily consumption of one dose (2 servings) of freeze-dried whole table grape powder, made from conventionally grown grapes to alter the composition of the bacteria that live in the intestines in healthy subjects. The grape powder contains 46g of individually quick frozen (IQF) grapes, which is equivalent to 252g fresh fruit. 20 subjects will will consume the beige diet for 4 weeks followed by one dose (two servings) of standardized Freeze-Dried Whole Table Grape Powder (46g) daily for 4 weeks. The primary objective of this pilot study is to determine changes in the gut microbiome. Stool samples will be collected at 4 and 8 weeks for bacterial DNA to determine changes in the bacteria that live in the intestines. You will be asked to avoid foods rich in polyphenols including dark chocolate and cocoa products, dried herbs, berries, coffee, tea, flaxseeds, nuts (chestnut, hazelnut), olive and artichoke for the duration of the study.

DETAILED DESCRIPTION:
The bacterial composition of the intestinal microbiome has been linked to the development of chronic diseases including obesity, metabolic syndrome, type II diabetes and heart disease. Grapes provide a rich source of polyphenols and fiber. It has been demonstrated in animal studies that fruits with high polyphenol content and fiber exhibit prebiotic effects leading to changes in the gut microbiome, decrease in symptoms of metabolic syndrome, improvement in insulin resistance and decrease in intestinal and systemic inflammation. Several human intervention studies have also been performed that demonstrated beneficial effects of high polyphenol fruits on the intestinal microbiome. No information is available about the effect of grape consumption on the gut microbiome. This proposed pilot study will assess the ability of consumption of two servings of grapes daily to alter the gut microbiome composition, leading to increased bile secretion, increased fecal cholesterol degradation/excretion, decreased plasma cholesterol and improved intestinal wellbeing in a free-living population. 20 subjects will consume the beige diet for 4 weeks followed by one dose (two servings) of standardized Freeze-Dried Whole Table Grape Powder (46g) daily for 4 weeks. The primary objective of this pilot study is to determine changes in the gut microbiome. Secondary outcome will be fecal bile and cholesterol and their metabolites, plasma cholesterol and intestinal wellbeing questionnaire at 4 and 8 weeks Stool samples will be collected at 4 and 8 weeks for sequencing of bacterial DNA to determine changes in the microbiota. Changes in fecal bile, cholesterol, and cholesterol metabolites will be analyzed by gas chromatography. The objective of the proposed pilot study is to determine whether intake of 2 servings of grapes per day will alter the intestinal microflora leading to an increase in intestinal cholesterol degradation, decreased plasma cholesterol and increased intestinal wellbeing. This project will provide novel preliminary data for future research studies and to develop new consumer messages on the gut health benefits of grapes. New consumer information about the health benefit of grapes will enhance the The California Table Grape industry domestic and export marketing programs and increase consumption of grapes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adults age 18-55 years old (females have to be premenopausal)
* Typically consume low fiber/polyphenol diet (beige diet)

Exclusion Criteria:

* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement, which interfere with the absorption of polyphenols.
* History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
* Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Is unable or unwilling to comply with the study protocol.
* Using prebiotics, probiotics, yogurt, and/or any fiber supplements regularly
* Allergy or sensitivity to grapes. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive affirmation by the subject of grape ingestion without incident will be requested.
* Taking antibiotics or laxatives within the past 3 months
* Allergy or sensitivity to grapes. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive history of grape ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
* Subjects with known allergy to food coloring dyes.
* In the opinion of the study investigator, any subject who demonstrate a risk of non-compliance with study procedure, or one who cannot read, understand or complete study - related materials.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in intestinal microbiome composition | Baseline (week 0) to Week 8
  Stool samples will be collected at week 4 and 8 of the intervention periods

SECONDARY OUTCOMES:
change in fecal cholesterol, cholesterol metabolites, and bile acids | Baseline (week 0) to Week 8
  Stool samples will be collected at week 4 and 8 of the intervention periods
change in blood total cholesterol, LDL and HDL-cholesterol, | Baseline (week 0) to Week 8
  Total cholesterol in blood will be analyzed spectrophotometrically using cholesterol reagent
digestive Health and General Wellness questionnaires (Rand SF-36) | Baseline (week 0) to Week 8
  The Weekly Digestive Symptom Log measures gastrointestinal symptoms (gas, bloating, diarrhea, etc.) and will be completed daily by all subjects. The Rand SF-36 will be completed at baseline (week 0), and week 4 visits to report on patients' overall well-being
urine content of syringic acid, and ellagic acid metabolites - ellagic acid, and dimethylellagic acid glucuronide | Baseline (week 0) to Week 8
  as biomarkers for compliance

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — UCLA Center for Human Nutrition
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No